CLINICAL TRIAL: NCT02741583
Title: Asthma Rehabilitation at High vs. Low Altitude: Randomized Controlled Parallel-group Trial
Brief Title: Kyrgyz Asthma Rehabilitation at High Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Req-2016-00076
Record Dates: First submitted 2016-04-12; First posted 2016-04-18 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Effect of High Altitude
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- altitude rehabilitation program (Experimental): 3 weeks rehabilitation program at high altitude (3200m)
  Interventions: Other: altitude rehabilitation program
- rehabilitation program (Active Comparator): 3 weeks rehabilitation program at low altitude (760m)
  Interventions: Other: rehabilitation program

INTERVENTIONS:
Other: altitude rehabilitation program — altitude exposure
  Arms: altitude rehabilitation program
Other: rehabilitation program — Rehabilitation at low altitude
  Arms: rehabilitation program

SUMMARY:
prospective controlled interventional trial evaluating the efficacy of a 3-weeks asthma rehabilitation program at high altitude (3200m) and low altitude (760m) on lung function and asthma control.

DETAILED DESCRIPTION:
Low altitude baseline measurements will be performed in Bishkek. Participants will then either be assigned to a rehabilitation program in Bishkek (760m) or in Tuja Ashu (3200m).

The rehabilitation programs in high or low altitude will be identically performed and will comprise

* asthma education and awareness
* instruction on inhaled therapies
* smoking cessation counseling
* respiratory and skeletal muscle training in groups
* guided walks / cycle ergometer training
* questionnaires on asthma control, quality of life
* spirometry and peak flow measurements
* echocardiography

Measurement on study subjects will be performed at baseline (Bishkek), during the rehabilitation program, after completion of the rehabilitation program and during a follow-up at week 15.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with atopic or non-atopic Asthma for at least 3 months
* partly controlled on regular or on demand inhaled therapy according to guidelines.
* asthma variability in peak expiratory flow > 10%/day and/or a reversible airflow obstruction in spirometry
* History of asthma consisting of variable symptoms (cough, dyspnea, wheezing).

Exclusion Criteria:

* Unstable and severely uncontrolled asthma needing systemic corticosteroids.
* Need of continuous oral steroids for their asthma control
* Heavy smokers (>20 cigarettes per day)
* Severe concomitant diseases preventing patients to adhere to the protocol and/or altitude exposure (severe metabolic, kidney- or liver disease, heart failure (ejection fracture <50%).
* Chronic lung diseases with a persistent FVC < 60% an/or arterial oxygen saturation <92%).
* Severe mental- or musculoskeletal disorders
* Pregnant or breast feeding women
* Patient which are unable to comply with the study procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
daily peak-flow variability | assessed at baseline, at run time of the rehabilitation program and 15 weeks after baseline measurements
change in asthma control questionnaire score | baseline to week 3 and 15

SECONDARY OUTCOMES:
forced expiratory volume in 1 second (FEV1) | baseline to week 3 and 15
average peak flow over 2 days | baseline to week 3 and 15
spirometric values (Forced vital capacity (FVC), FEV1/FVC) | from baseline to week 3 and 15
asthma-related quality of life (AQLQ) | from baseline to week 3 and 15
generic quality of life (Short-Form 36(SF-36)) | from baseline to week 3 and 15
symptoms of acute mountain sickness (AMS) by the environmental symptom cerebral score (AMS-c) | from baseline to week 3 and 15
6 minute walk distance | from baseline to week 3 and 15
sit-to-stand test | from baseline to week 3 and 15
arterial oxygen saturation by pulse oximetry | from baseline to week 3 and 15
visual analog scale (VAS) | from baseline to week 3 and 15

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich Somaini, MD, Study Chair — University of Zurich
Locations (1):
- Respiratory Clinic, University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Saxer S, Schneider SR, Appenzeller P, Bader PR, Lichtblau M, Furian M, Sheraliev U, Estebesova B, Emilov B, Sooronbaev T, Bloch KE, Ulrich S. Asthma rehabilitation at high vs. low altitude: randomized parallel-group trial. BMC Pulm Med. 2019 Jul 24;19(1):134. doi: 10.1186/s12890-019-0890-y. PMID 31340793